CLINICAL TRIAL: NCT03516383
Title: Pulse Wave Velocity Imaging in the Assessment of PAD
Acronym: PWVi
Status: Withdrawn | Type: Observational
Why Stopped: No funding received.
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-028
Record Dates: First submitted 2016-05-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: PAD; Optical Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: * ABI < 0.6, confirmed PAD
  * 50 - 90 years of age
  * In-patients or out-patients
  * Participants who understand the study and are able to give consent
  * Participants who can be followed by the same investigating team for the whole period of their participation in the study
  Interventions: Device: PWVi
- Control: * ABI of 0.9 < ABI < 1.2
  * 50 - 90 years of age
  * Participants who understand the study and are able to give consent
  * Participants who can be followed by the same investigating team for the whole period of their participation in the study
  Interventions: Device: PWVi

INTERVENTIONS:
Device: PWVi

SUMMARY:
The purpose of this study is to predict the outcome of peripheral revascularization surgery by use of a new technology developed by our team, Pulse Wave Velocity imaging (PWVI), which has the capability to detect pulse transit time (PTT), and pulse wave velocity (PWV). This PWVI will be compared against known gold standards pre and post lower extremity limb revascularization and used to evaluate outcomes. Specifically, is leg PWV different among those with or without PAD, and is leg PWV different among those who undergo revascularization surgery and those who do not? This study represents the first clinical pilot study of the device with the aim to expand study participant numbers in future research and to eventually develop a PAD screening tool. This would be the first of its kind ever described.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is the narrowing of arteries in the extremities, resulting in insufficient blood supply to tissue in the extremities. In its mildest form, PAD may be asymptomatic, or may show mild symptoms such as intermittent claudication (IC), a pain one may experience while walking. [Hirsch et al, 2006; Criqui et al, 1992; Beckman, 2002] At its extreme, PAD may lead to critical limb ischaemia (CLI), necrosis, gangrene, amputation, or even death. [Hirsch et al, 2006; Hirsch et al, 2001; Criqui et al, 1992] PAD affects over 20% of all patients aged 70 and above, or aged 50 to 69 with a history of smoking or diabetes. [Hirsch et al, 2001; Beckman et al, 2006] In primary care, the ankle-brachial index (ABI) has been used as a screening tool for PAD. [Aboyans et al., 2012] The ABI consists of the ratio of systolic blood pressures measured at the ankle to that of the brachial artery. An ABI of 0.9 - 1.1 is considered normal, and ABI ≤ 0.9 is considered abnormal. [Aboyans et al., 2012; Hirsch et al., 2001] By way of the ABI, a primary care practitioner may be able to diagnose PAD with a high degree of specificity (up to 99%), but sensitivity can vary greatly (15-79%). [Xu et al, 2010] More recently, the use of the brachial-ankle pulse wave velocity (baPWV) has been used as another diagnostic tool with regards to coronary artery disease (CAD). [Katakami et al., 2014; Chae et al., 2013; Yamashina et al., 2002] Sugawara et al. have shown that the variability in the baPWV is due 58% to aortic pulse wave velocity (PWV), and 23% to leg PWV. [Sugawara et al., 2005] Although aortic stiffness is a larger component of the baPWV, numerous studies have shown that there is a correlation between baPWV and PAD. [Yokoyama et al., 2003; Amoh-Tonto et al., 2009; Xu et al., 2008] Additionally, it has been shown that baPWV can increase after percutaneous transluminal angioplasty in the lower extremities. [Yokoyama et al., 2003] In context with CLI, although methods of diagnosis have improved over the past decades, amputation rates have seen an increase. [Beckman, 2007] Revascularization surgery has been shown to increase ambulatory function and quality of life in those affected by CLI as compared to those who had undergone amputation. [Brosi et al., 2007; Deneuville & Perrouillet, 2006; Oresanya et al, 2015] This, and the cut-off ABI value <0.95 set by Motobe et al. in 2005 for the accuracy of baPWV measurements, requires further investigation into leg PWV for a better understanding of PAD and CLI and the effects revascularization surgery has. [Wohlfart et al., 2013] The investigators believe that the ability to determine the success of revascularization surgery at the time of surgery would guide vascular surgeons in the intra-operative treatment and monitoring of these patients. The current standard of care is Doppler of the dorsalis pedis or posterior tibial artery post-operatively and at the bedside. This is not always an accurate determinate of the success of a revascularized limb and subsequently patients require either Duplex ultrasound, computed tomography angiography (CTA) or angiography. The results from these more sophisticated investigations provide accurate information about blood flow and its characteristics. Our group has designed a device called Pulse Wave Velocity imaging (PWVI). This device has the capacity to determine pulse wave velocity, pulse transit time and a waveform analysis at the bedside and can be designed as a small handheld tool. This is essentially a culmination of the information obtained from Duplex ultrasound and photoplethysmography but can be acquired within 30 seconds in any environment (eg. Operating room, bedside, patient's home).

ELIGIBILITY:
Inclusion Criteria Group 1. Control (n=10)

* ABI of 0.9 < ABI < 1.2
* 50 - 90 years of age
* Participants who understand the study and are able to give consent
* Participants who can be followed by the same investigating team for the whole period of their participation in the study Group 2. Experimental (n=10)
* ABI < 0.6, confirmed PAD
* 50 - 90 years of age
* In-patients or out-patients
* Participants who understand the study and are able to give consent
* Participants who can be followed by the same investigating team for the whole period of their participation in the study

Exclusion Criteria Group 1. Control (n=10)

* Diabetics
* Smokers
* Body mass index (BMI) > 35 Group 2. Experimental (n=10)
* Diabetics
* Smokers
* Advanced lymphedema or dermatoliposclerosis
* BMI > 35

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1 (n=10), the control group, will be recruited via referral from our research team and will consist of healthy individuals with a normal ABI of 0.9 < ABI < 1.2. Group 2 (n=10), participants with PAD, ABI < 0.6, either requiring revascularization surgery (group 2B, n=5), or not (group 2A, n=5). These participants will be recruited from the population routinely seen by the Principal Investigators or team members.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Waveform Imaging using Pulse Wave Velocity | 8 weeks
  Using new technology to measure tissue viability in surgical participants.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cross, MD, PhD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Background] Beckman JA, Jaff MR, Creager MA. The United States preventive services task force recommendation statement on screening for peripheral arterial disease: more harm than benefit? Circulation. 2006 Aug 22;114(8):861-6. doi: 10.1161/CIRCULATIONAHA.105.607846. PMID 16923770